CLINICAL TRIAL: NCT06160037
Title: Influence of Prenatal and Early Childhood Home-Visiting by Nurses on Development of Chronic Disease: 29-year Follow-Up of a Randomized Clinical Trial
Brief Title: Influence of Prenatal and Early Childhood Home-Visiting by Nurses on Development of Chronic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Rochester (Other); Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-0794
Record Dates: First submitted 2023-11-14; First posted 2023-12-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease | interventions — Transportation; Mass Screening

STUDY DESIGN:
Intervention Model Description: Longitudinal cohort study
Who Masked: Outcomes Assessor
Masking Description: Those involved in conducting assessments of study participants have been masked to treatment assignment for the 30-year period following study enrollment during pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1. Transportation and Screening (Active Comparator): Free transportation for scheduled prenatal care, developmental screening and referral services for the child at the 6th, 12th, and 24th months of the child's life.
  Interventions: Behavioral: Transportation and Developmental Screening
- Arm 2. Transportation, Screening, and Nurse-Visitation during Pregnancy and Infancy (Experimental): Free transportation for scheduled prenatal care; intensive nurse home-visitation services during pregnancy and through the child's second birthday; and developmental screening and referral services for the child at the 6th, 12th, and 24th months of the child's life.
  Interventions: Behavioral: Transportation, Screening, and Nurse-Visitation during Pregnancy and Infancy

INTERVENTIONS:
Behavioral: Transportation and Developmental Screening — Arm 1. Transportation and Screening The 514 families in this condition received: 1) free transportation for scheduled prenatal care; and 2) developmental screening and referral services for the child at the 6th, 12th, and 24th months of the child's life.
  Arms: Arm 1. Transportation and Screening
Behavioral: Transportation, Screening, and Nurse-Visitation during Pregnancy and Infancy — Arm 2. Transportation, Screening, and Nurse-Visitiation During Pregnancy and Infancy
  The 228 families in this condition received: 1) free transportation for scheduled prenatal care; 2) intensive nurse home-visitation services during pregnancy and through the child's second birthday; and 3) developmental screening and referral services for the child at the 6th, 12th, and 24th months of the child's life.
  Arms: Arm 2. Transportation, Screening, and Nurse-Visitation during Pregnancy and Infancy

SUMMARY:
This study is a longitudinal cohort study that follows participants in a randomized clinical trial of a program of prenatal and early child home visiting on maternal and offspring risks for chronic disease.

DETAILED DESCRIPTION:
Addressing the unacceptably high rates of chronic disease and premature mortality among low-income African Americans (AA) is a public health imperative. The proposed study addresses this challenge by building upon decades of follow-up of low-income, primarily AA participants in a randomized clinical trial of the Nurse-Family Partnership (NFP), a program of prenatal and infant/toddler nurse home visiting for low-income mothers with no previous live births. It examines NFP effects on risks for cardiovascular disease (CVD), type 2 diabetes (T2D), and chronic kidney disease (CKD), as well as premature mortality among both mothers and their first-born offspring at offspring age 30. It is the first adequately powered study of a very early intervention to examine risks for chronic disease and mortality, assessing both mothers and their first-born offspring.

Please note that for this section of the longitudinal study, just the outcome measures for 30 years after delivery are being measured. The study team also measured these outcome measures at baselines, 12 years, and 18 years after delivery in other studies, but for this specific study, the time frame for the listed outcome measures is 30 years after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who participated in a randomized clinical trial of nurse home visiting and their first-born offspring.
* Women < 29 weeks pregnant --> No previous live births
* No specific chronic illnesses thought to contribute to fetal growth retardation or preterm delivery
* At least two of the following sociodemographic risk conditions: unmarried, less than 12 years of education, and unemployed

Exclusion Criteria:

* Participants who refused assessments at earlier phases of data gathering.
* Women > 29 weeks pregnant
* Previous live births
* Possessing chronic illnesses like hypertensive disorders requiring medical treatment, severe cardiac disease, large uterine fibroids.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1055 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Height (standing) | Approximately 30 years after delivery
  Description: height measured in cm while participant is standing in bare feet using a stationary stadiometer with headpiece
Weight | Approximately 30 years after delivery
  weight measured in pounds
Waist circumference | once, approximately 30 years after delivery.
  waist circumference measured in cm, after exhaling, just above iliac crest, using a non-stretchable cloth measuring tape.
Hip circumference | once, approximately 30 years after delivery
  hip circumference measured in cm, at point of greatest protrusion of gluteal muscles, using a non-stretchable cloth.
Percent total body fat | once, approximately 30 years after delivery
  Measured using the Tanita-780U Multifrequency Segmental Body Composition Analyzer
% body fat in arms, legs | once, approximately 30 years after delivery
  Measured using the Tanita-780U Multifrequency Segmental Body Composition Analyzer
Visceral (trunk) fat | once, approximately 30 years after delivery
  Measured using the Tanita-780U Multifrequency Segmental Body Composition Analyzer
Total Cholesterol (TC), High density lipoprotein (HDL), Low density lipoprotein (LDL) | once, approximately 30 years after delivery
  TC, HDL, and LDL are measured by a clinical laboratory from serum samples by Medpace Laboratories.
Triglycerides | once, approximately 30 years after delivery
  Measured by a clinical laboratory from serum samples by Medpace Laboratories
Glycosylated hemoglobin | once, approximately 30 years after delivery
  Measured by a clinical laboratory from whole blood samples by Medpace Laboratories
Insulin-like growth factor 1 (IGF-1) | once, approximately 30 years after delivery
  IGF-1 is a hormonal mediator and is analyzed in serum by Medpace Laboratories.
Follicle-Stimulating Hormone (FSH) | once, approximately 30 years after delivery
  FSH is an indicator of menopausal status and is measured in serum by the Medpace Laboratories.
Urine-Albumin | once, approximately 30 years after delivery
  URINE albumin is measured by Medpace Laboratories
Urine Creatinine | once, approximately 30 years after delivery
  Urine creatinine is measured in urine by Medpace Laboratories.
Estimated Glomerular Filtration Rate (eGFR) | once, approximately 30 years after delivery
  eGFR (estimated glomerular filtration rate) is calculated based on serum creatinine value, age, and gender; measured by Medpace Laboratories.
High sensitivity C-reactive protein (hs CRP) | once, approximately 30 years after delivery
  hs-CRP measured in plasma by Medpace Laboratories . This is an inflammatory marker.
Interleukin-6 (IL-6) | once, approximately 30 years after delivery
  IL-6 measured in serum by Medpace laboratory. This is an inflammatory marker.
Tumor Necrosis Factor alpha receptor 2 | once, approximately 30 years after delivery
  Tumor Necrosis Factor alpha receptor 2 (TNF alpha receptor 2) is measured in serum by Medpace Laboratories. This is an inflammatory marker.
Fibrinogen | once, approximately 30 years after delivery
  Fibrinogen is measured in plasma by Medpace Laboratories. This is an inflammatory marker.
Resting blood pressure (diastolic) | once, approximately 30 years after delivery
  Blood pressure read measured through SphygmoCor XCEL, taken after 10 minutes of sitting quietly.
Resting blood pressure (systolic) | once, approximately 30 years after delivery
  Blood pressure read measured through SphygmoCor XCEL, taken after 10 minutes of sitting quietly.
Carotid to femoral pulse wave velocity (cf-PWV) | once, approximately 30 years after delivery
  Pulse wave velocity is a measure of arterial stiffness. It is a predictor of cardiovascular risk. It is measured using the SphygmoCor XCEL instrument.
Augmentation index | once, approximately 30 years after delivery
  Augmentation Index is a measure of arterial stiffness. It is calculated as the ratio of Augmented Pressure to Pulse pressure. a predictor of cardiovascular risk. It is measured using the SphygmoCor SCEL instrument
Mortality - Mothers | measured once, approximately 30 years after delivery.
  The study team expects the intervention to reduce the rates of all-cause mortality among mothers given that death is more likely among those with COVID infections who have underlying chronic conditions. Moreover, the study team expects the program to reduce mortality for chronic diseases and CVD among mothers if the rates are sufficiently high to detect such differences.
Mortality - Offspring | measured once, approximately 30 years after delivery.
  Among offspring, those who become infected with COVID are less likely to die than their mothers, given that their underlying chronic conditions are less likely to be as serious or prevalent. Therefore, the investigators expect the treatment-control differences to be limited to external causes.
  Note that in the original proposal the authors had included deaths due preventable causes (SIDS) as operationalized in a recent publication: https://pubmed.ncbi.nlm.nih.gov/34420828/. Given the controversy that has emerged in recent years about whether the causes of SIDS are uniformly preventable, SIDS was added to a modified version of this outcome that includes external cuases, that will be analyzed as an exploratory outcome in examining offspring mortality. The authors also will conduct an exploratory analysis of all-cause mortality.

SECONDARY OUTCOMES:
Medical diagnoses, signs, and symptoms | interview conducted approximately 30 years after delivery
  Obtained via medical history interview by trained nurses.
Current medications | interview conducted approximately 30 years after delivery
  Obtained via medical history interview by trained nurses.
Number of Hospitalizations per participant (mental/behavioral) | interview conducted approximately 30 years after delivery
  Obtained via medical history interview by trained nurses, and by matching administrative hospitalization records (in Tennessee only) to study subjects who have given consent.
Number of Hospitalizations per participant (medical/surgical) | interview conducted approximately 30 years after delivery
  Obtained via medical history interview by trained nurses, and by matching administrative hospitalization records (in Tennessee only) to study subjects who have given consent.
Disability (injury) | interview conducted approximately 30 years after delivery
  obtained from 1) administrative data on Social Security disability payment and 2) information derived from the interview regarding if and why participant is receiving Supplemental Security Income.
Disability (physical) | interview conducted approximately 30 years after delivery
  1) administrative data on Social Security disability payment and 2) information derived from the interview regarding if and why participant is receiving Supplemental Security.
Disability (mental illness) | interview conducted approximately 30 years after delivery
  1) administrative data on Social Security disability payment and 2) information derived from the interview regarding if and why participant is receiving Supplemental Security Income.
Number of pregnancies | interview conducted approximately 30 years after delivery
  Self-reports of all pregnancies and dates
Pregnancy losses | interview conducted approximately 30 years after delivery
  self-reports of all pregnancies not resulting in a live birth
Number of live births | interview conducted approximately 30 years after delivery
  1) self-reports of all children's dates of births and 2) administrative data
Pregnancy complications | interview conducted approximately 30 years after delivery
  derived from administrative (birth certificate) data
Birthweight | interview conducted approximately 30 years after delivery
  determined through a combination of interview and administrative (birth certificate) data
Gestational age | interview conducted approximately 30 years after delivery
  determined through a combination of interview and administrative (birth certificate) data
Menopause (age) | interview conducted approximately 30 years after delivery
  Determined via interview
Self-rated health | interview conducted approximately 30 years after delivery
  Excellent, very good, good, fair, or poor
Physical activity - Total Metabolic Equivalent of Task (MET) minutes per week | interview conducted approximately 30 years after delivery
  International Physical Activity Questionnaire (IPAQ): questionnaire to obtain internationally comparable data regarding physical activity. Questions ask about quantity and duration of physical activity.
Sleep Quality -- Global Score | interview conducted approximately 30 years after delivery
  Derived from Pittsburgh Sleep Quality Index (PSQI): questions on the PSQI are rated on a scale of 0-3, 0 = no difficulty to 3 = severe difficulty, and ask questions related to sleep latency, sleep duration, sleep disturbances, use of sleep medication,and daytime dysfunction.
Average daily fruit and vegetable intake | interview conducted approximately 30 years after delivery
  derived from Diet NIH Eating at America's Table: All-Day Fruit & vegetable Screener
Percent energy from fat | interview conducted approximately 30 years after delivery
  Derived from National Cancer Institute Percentage Energy from Fat Screener
Dietary restraint/eating patterns | interview conducted approximately 30 years after delivery
  Derived from Three Factor Eating Questionnaire: Measures three aspects of eating behaviors: cognitive restraint, uncontrolled eating, and emotional eating.
Screening for Substance Use - TAPS 1 (tobacco, alcohol, prescription medication, and other substance use) | interview conducted approximately 30 years after delivery
  use of substances in the past three months
Substance Use Risk Level TAPS 2 | interview conducted approximately 30 years after delivery
  Risk category: no use in past 3 months, problem use, higher risk Substance Use Dependence
Tobacco: Cigarettes | interview conducted approximately 30 years after delivery
  Ever smoked cigarettes, age started and stopped smoking, number of cigarettes per day
Tobacco: Cigars | interview conducted approximately 30 years after delivery
  Ever smoked cigars, aged started and stopped, number of cigars per week
Tobacco: Pipe, Hookah | interview conducted approximately 30 years after delivery
  Ever smoke tobacco in pipe or hookah, age started and stopped, number of pipe bowls per week
Tobacco: Smokeless Tobacco Snus | interview conducted approximately 30 years after delivery
  Ever used Snus, age started and stopped, number of snus pouches per week
Other Smokeless Tobacco (dip, chewing tobacco) | interview conducted approximately 30 years after delivery
  : Ever used dip, chewing tobacco, age started and stopped, number of times per day
Tobacco: Electronic Nicotine Products | interview conducted approximately 30 years after delivery
  Ever used, age started and stopped, number of times per day
Depression | interview conducted approximately 30 years after delivery
  Derived from the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression 8a Adult: measures patient-reported outcomes like pain, fatigue, physical functioning, emotional distress, and social role participation.Each question uses a 5-point ordinal scale of "never," "rarely," sometimes," "often," and "always." Higher scores indicate higher depression severity.
Anxiety | interview conducted approximately 30 years after delivery
  Derived from the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety 8a Adult. 7 Questions about feelings related to anxiety felt in the past seven days. Each question uses a 5-point ordinal scale of "never," "rarely," sometimes," "often," and "always." Higher scores indicate higher anxiety severity.
Mastery | interview conducted approximately 30 years after delivery
  Derived from Pearlin Mastery Scale. Measured on a 4 point Likert Scale, (1: Strongly Disagree, 4: Strongly agree). Scores can range from 7-28, with higher scores indicating a higher level of mastery.
Duration of Marriage and partnered relationships | interview conducted approximately 30 years after delivery
  List of current and previous married and partnered relationships, length of time together.
Relationship Commitment: Current Relationship | interview conducted approximately 30 years after delivery
  Structural commitment (dating, cohabitating, married)
Relationship Personal Commitment: Current Relationship | interview conducted approximately 30 years after delivery
  not at all committed to extremely committed relationship: 2 indicators of committment: structural and personal commitment. Personal commitment responses: 1-4, 1: not very committed, to 4: extremely committed.
Relationship Satisfaction: Current Relationship | interview conducted approximately 30 years after delivery
  Overall happiness with relationship and satisfaction with partner: assessed with 2 questions regarding overall happiness and partner satisfaction.
Partner Warmth Index: Current Relationship | interview conducted approximately 30 years after delivery
  Degree to which partner displayed warm behaviors: 3 questions regarding how often their partner displayed warm behaviors in the past month, ranging from 1-4. 1: never to 4: always.
Partner Hostility Index: Current Relationship | interview conducted approximately 30 years after delivery
  Degree to which partner displayed hostile behaviors: 5 questions asking about partner hostile behavior in past month, ranging from 1-4. 1: never, 4: always
Educational attainment (High School) | interview conducted approximately 30 years after delivery
  High school education: graduated from high school, obtained General Education Development (GED), left high school without completing.
Educational attainment (College) | interview conducted approximately 30 years after delivery
  Highest Degree completed: Associates, Bachelors, Masters, PhD.
Educational attainment (job training) | interview conducted approximately 30 years after delivery
  Dates and types of job training programs
Current work status (job) | interview conducted approximately 30 years after delivery
  List of employment, duties, dates of employment
Current work status (hours/week) | interview conducted approximately 30 years after delivery
  number of hours work per week
Arrests and Incarceration | interview conducted approximately 30 years after delivery
  Dates and outcomes of arrests
Arrests | interview conducted approximately 30 years after delivery
  Types of arrests: misdemeanor, felony
Arrests and incarceration | interview conducted approximately 30 years after delivery
  number of days incarcerated

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators are only sharing IPD among the institutions involved in the conduct of this study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: March 1, 2025
Access Criteria: check with Nancy about this

REFERENCES:
- [Background] Carnethon MR, Pu J, Howard G, Albert MA, Anderson CAM, Bertoni AG, Mujahid MS, Palaniappan L, Taylor HA Jr, Willis M, Yancy CW; American Heart Association Council on Epidemiology and Prevention; Council on Cardiovascular Disease in the Young; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Functional Genomics and Translational Biology; and Stroke Council. Cardiovascular Health in African Americans: A Scientific Statement From the American Heart Association. Circulation. 2017 Nov 21;136(21):e393-e423. doi: 10.1161/CIR.0000000000000534. Epub 2017 Oct 23. PMID 29061565
- [Background] Cunningham TJ, Croft JB, Liu Y, Lu H, Eke PI, Giles WH. Vital Signs: Racial Disparities in Age-Specific Mortality Among Blacks or African Americans - United States, 1999-2015. MMWR Morb Mortal Wkly Rep. 2017 May 5;66(17):444-456. doi: 10.15585/mmwr.mm6617e1. PMID 28472021
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Menke A, Casagrande S, Geiss L, Cowie CC. Prevalence of and Trends in Diabetes Among Adults in the United States, 1988-2012. JAMA. 2015 Sep 8;314(10):1021-9. doi: 10.1001/jama.2015.10029. PMID 26348752
- [Background] United States Renal Data System. 2014 USRDS annual data report: Epidemiology of kidney disease in the United States. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases: Bethesda, MD, 2014.
- [Background] Havranek EP, Mujahid MS, Barr DA, Blair IV, Cohen MS, Cruz-Flores S, Davey-Smith G, Dennison-Himmelfarb CR, Lauer MS, Lockwood DW, Rosal M, Yancy CW; American Heart Association Council on Quality of Care and Outcomes Research, Council on Epidemiology and Prevention, Council on Cardiovascular and Stroke Nursing, Council on Lifestyle and Cardiometabolic Health, and Stroke Council. Social Determinants of Risk and Outcomes for Cardiovascular Disease: A Scientific Statement From the American Heart Association. Circulation. 2015 Sep 1;132(9):873-98. doi: 10.1161/CIR.0000000000000228. Epub 2015 Aug 3. No abstract available. PMID 26240271
- [Background] Pool LR, Ning H, Lloyd-Jones DM, Allen NB. Trends in Racial/Ethnic Disparities in Cardiovascular Health Among US Adults From 1999-2012. J Am Heart Assoc. 2017 Sep 22;6(9):e006027. doi: 10.1161/JAHA.117.006027. PMID 28939713
- [Background] Bancks MP, Kershaw K, Carson AP, Gordon-Larsen P, Schreiner PJ, Carnethon MR. Association of Modifiable Risk Factors in Young Adulthood With Racial Disparity in Incident Type 2 Diabetes During Middle Adulthood. JAMA. 2017 Dec 26;318(24):2457-2465. doi: 10.1001/jama.2017.19546. PMID 29279935
- [Background] Signorello LB, Schlundt DG, Cohen SS, Steinwandel MD, Buchowski MS, McLaughlin JK, Hargreaves MK, Blot WJ. Comparing diabetes prevalence between African Americans and Whites of similar socioeconomic status. Am J Public Health. 2007 Dec;97(12):2260-7. doi: 10.2105/AJPH.2006.094482. Epub 2007 Oct 30. PMID 17971557
- [Background] Norton JM, Moxey-Mims MM, Eggers PW, Narva AS, Star RA, Kimmel PL, Rodgers GP. Social Determinants of Racial Disparities in CKD. J Am Soc Nephrol. 2016 Sep;27(9):2576-95. doi: 10.1681/ASN.2016010027. Epub 2016 May 13. PMID 27178804
- [Background] Stuart-Shor EM, Berra KA, Kamau MW, Kumanyika SK. Behavioral strategies for cardiovascular risk reduction in diverse and underserved racial/ethnic groups. Circulation. 2012 Jan 3;125(1):171-84. doi: 10.1161/CIRCULATIONAHA.110.968495. No abstract available. PMID 22215892
- [Background] Suglia SF, Koenen KC, Boynton-Jarrett R, Chan PS, Clark CJ, Danese A, Faith MS, Goldstein BI, Hayman LL, Isasi CR, Pratt CA, Slopen N, Sumner JA, Turer A, Turer CB, Zachariah JP; American Heart Association Council on Epidemiology and Prevention; Council on Cardiovascular Disease in the Young; Council on Functional Genomics and Translational Biology; Council on Cardiovascular and Stroke Nursing; and Council on Quality of Care and Outcomes Research. Childhood and Adolescent Adversity and Cardiometabolic Outcomes: A Scientific Statement From the American Heart Association. Circulation. 2018 Jan 30;137(5):e15-e28. doi: 10.1161/CIR.0000000000000536. Epub 2017 Dec 18. PMID 29254928
- [Background] Slopen N, Loucks EB, Appleton AA, Kawachi I, Kubzansky LD, Non AL, Buka S, Gilman SE. Early origins of inflammation: An examination of prenatal and childhood social adversity in a prospective cohort study. Psychoneuroendocrinology. 2015 Jan;51:403-13. doi: 10.1016/j.psyneuen.2014.10.016. Epub 2014 Oct 25. PMID 25462912
- [Background] Loria AS, Ho DH, Pollock JS. A mechanistic look at the effects of adversity early in life on cardiovascular disease risk during adulthood. Acta Physiol (Oxf). 2014 Feb;210(2):277-87. doi: 10.1111/apha.12189. Epub 2013 Dec 13. PMID 24330084
- [Background] Alexander BT, Dasinger JH, Intapad S. Fetal programming and cardiovascular pathology. Compr Physiol. 2015 Apr;5(2):997-1025. doi: 10.1002/cphy.c140036. PMID 25880521
- [Background] Mor G, Cardenas I. The immune system in pregnancy: a unique complexity. Am J Reprod Immunol. 2010 Jun;63(6):425-33. doi: 10.1111/j.1600-0897.2010.00836.x. Epub 2010 Mar 29. PMID 20367629
- [Background] Brunton PJ, Russell JA. Endocrine induced changes in brain function during pregnancy. Brain Res. 2010 Dec 10;1364:198-215. doi: 10.1016/j.brainres.2010.09.062. Epub 2010 Sep 22. PMID 20869351
- [Background] Fisher C, MacLean M, Morecroft I, Seed A, Johnston F, Hillier C, McMurray J. Is the pregnancy hormone relaxin also a vasodilator peptide secreted by the heart? Circulation. 2002 Jul 16;106(3):292-5. doi: 10.1161/01.cir.0000025630.05387.45. PMID 12119241
- [Background] Sanghavi M, Rutherford JD. Cardiovascular physiology of pregnancy. Circulation. 2014 Sep 16;130(12):1003-8. doi: 10.1161/CIRCULATIONAHA.114.009029. No abstract available. PMID 25223771
- [Background] Hoekzema E, Barba-Muller E, Pozzobon C, Picado M, Lucco F, Garcia-Garcia D, Soliva JC, Tobena A, Desco M, Crone EA, Ballesteros A, Carmona S, Vilarroya O. Pregnancy leads to long-lasting changes in human brain structure. Nat Neurosci. 2017 Feb;20(2):287-296. doi: 10.1038/nn.4458. Epub 2016 Dec 19. PMID 27991897
- [Background] Swain JE, Kim P, Spicer J, Ho SS, Dayton CJ, Elmadih A, Abel KM. Approaching the biology of human parental attachment: brain imaging, oxytocin and coordinated assessments of mothers and fathers. Brain Res. 2014 Sep 11;1580:78-101. doi: 10.1016/j.brainres.2014.03.007. Epub 2014 Mar 15. PMID 24637261
- [Background] Faraji J, Karimi M, Soltanpour N, Rouhzadeh Z, Roudaki S, Hosseini SA, Jafari SY, Abdollahi AA, Soltanpour N, Moeeini R, Metz GAS. Intergenerational Sex-Specific Transmission of Maternal Social Experience. Sci Rep. 2018 Jul 12;8(1):10529. doi: 10.1038/s41598-018-28729-8. PMID 30002484
- [Background] Wan L, Tu T, Zhang QL, Jiang J, Yan XX. Pregnancy Promotes Maternal Hippocampal Neurogenesis in Guinea Pigs. Neural Plast. 2019 Apr 11;2019:5765284. doi: 10.1155/2019/5765284. eCollection 2019. PMID 31097956
- [Background] Barba-Muller E, Craddock S, Carmona S, Hoekzema E. Brain plasticity in pregnancy and the postpartum period: links to maternal caregiving and mental health. Arch Womens Ment Health. 2019 Apr;22(2):289-299. doi: 10.1007/s00737-018-0889-z. Epub 2018 Jul 14. PMID 30008085
- [Background] Zhang S, Ding Z, Liu H, Chen Z, Wu J, Zhang Y, Yu Y. Association between mental stress and gestational hypertension/preeclampsia: a meta-analysis. Obstet Gynecol Surv. 2013 Dec;68(12):825-34. doi: 10.1097/OGX.0000000000000001. PMID 25102019
- [Background] Ying W, Catov JM, Ouyang P. Hypertensive Disorders of Pregnancy and Future Maternal Cardiovascular Risk. J Am Heart Assoc. 2018 Sep 4;7(17):e009382. doi: 10.1161/JAHA.118.009382. No abstract available. PMID 30371154
- [Background] Bergen NE, Schalekamp-Timmermans S, Roos-Hesselink J, Roeters van Lennep JE, Jaddoe VVW, Steegers EAP. Hypertensive disorders of pregnancy and subsequent maternal cardiovascular health. Eur J Epidemiol. 2018 Aug;33(8):763-771. doi: 10.1007/s10654-018-0400-1. Epub 2018 May 19. PMID 29779204
- [Background] Grandi SM, Filion KB, Yoon S, Ayele HT, Doyle CM, Hutcheon JA, Smith GN, Gore GC, Ray JG, Nerenberg K, Platt RW. Cardiovascular Disease-Related Morbidity and Mortality in Women With a History of Pregnancy Complications. Circulation. 2019 Feb 19;139(8):1069-1079. doi: 10.1161/CIRCULATIONAHA.118.036748. Erratum In: Circulation. 2019 Aug 27;140(9):e544. doi: 10.1161/CIR.0000000000000718. PMID 30779636
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams DJ. Pre-eclampsia and risk of cardiovascular disease and cancer in later life: systematic review and meta-analysis. BMJ. 2007 Nov 10;335(7627):974. doi: 10.1136/bmj.39335.385301.BE. Epub 2007 Nov 1. PMID 17975258
- [Background] Behrens I, Basit S, Melbye M, Lykke JA, Wohlfahrt J, Bundgaard H, Thilaganathan B, Boyd HA. Risk of post-pregnancy hypertension in women with a history of hypertensive disorders of pregnancy: nationwide cohort study. BMJ. 2017 Jul 12;358:j3078. doi: 10.1136/bmj.j3078. PMID 28701333
- [Background] Xu J, Barinas-Mitchell E, Kuller LH, Youk AO, Catov JM. Maternal hypertension after a low-birth-weight delivery differs by race/ethnicity: evidence from the National Health and Nutrition Examination Survey (NHANES) 1999-2006. PLoS One. 2014 Aug 5;9(8):e104149. doi: 10.1371/journal.pone.0104149. eCollection 2014. PMID 25093324
- [Background] Mamun AA, O'Callaghan MJ, Williams GM, Najman JM. Maternal smoking during pregnancy predicts adult offspring cardiovascular risk factors - evidence from a community-based large birth cohort study. PLoS One. 2012;7(7):e41106. doi: 10.1371/journal.pone.0041106. Epub 2012 Jul 19. PMID 22829913
- [Background] Gaillard R. Maternal obesity during pregnancy and cardiovascular development and disease in the offspring. Eur J Epidemiol. 2015 Nov;30(11):1141-52. doi: 10.1007/s10654-015-0085-7. Epub 2015 Sep 16. PMID 26377700
- [Background] Mamun AA, Kinarivala MK, O'Callaghan M, Williams G, Najman J, Callaway L. Does hypertensive disorder of pregnancy predict offspring blood pressure at 21 years? Evidence from a birth cohort study. J Hum Hypertens. 2012 May;26(5):288-94. doi: 10.1038/jhh.2011.35. Epub 2011 Apr 21. PMID 21509041
- [Background] Kajantie E, Eriksson JG, Osmond C, Thornburg K, Barker DJ. Pre-eclampsia is associated with increased risk of stroke in the adult offspring: the Helsinki birth cohort study. Stroke. 2009 Apr;40(4):1176-80. doi: 10.1161/STROKEAHA.108.538025. Epub 2009 Mar 5. PMID 19265049
- [Background] Smith CJ, Ryckman KK, Barnabei VM, Howard BV, Isasi CR, Sarto GE, Tom SE, Van Horn LV, Wallace RB, Robinson JG. The impact of birth weight on cardiovascular disease risk in the Women's Health Initiative. Nutr Metab Cardiovasc Dis. 2016 Mar;26(3):239-45. doi: 10.1016/j.numecd.2015.10.015. Epub 2015 Nov 18. PMID 26708645
- [Background] Doom JR, Mason SM, Suglia SF, Clark CJ. Pathways between childhood/adolescent adversity, adolescent socioeconomic status, and long-term cardiovascular disease risk in young adulthood. Soc Sci Med. 2017 Sep;188:166-175. doi: 10.1016/j.socscimed.2017.06.044. Epub 2017 Jul 24. PMID 28747248
- [Background] Gebreab SY, Diez Roux AV, Brenner AB, Hickson DA, Sims M, Subramanyam M, Griswold ME, Wyatt SB, James SA. The impact of lifecourse socioeconomic position on cardiovascular disease events in African Americans: the Jackson Heart Study. J Am Heart Assoc. 2015 May 27;4(6):e001553. doi: 10.1161/JAHA.114.001553. PMID 26019130
- [Background] Danese A, Moffitt TE, Harrington H, Milne BJ, Polanczyk G, Pariante CM, Poulton R, Caspi A. Adverse childhood experiences and adult risk factors for age-related disease: depression, inflammation, and clustering of metabolic risk markers. Arch Pediatr Adolesc Med. 2009 Dec;163(12):1135-43. doi: 10.1001/archpediatrics.2009.214. PMID 19996051
- [Background] Suglia SF, Clark CJ, Boynton-Jarrett R, Kressin NR, Koenen KC. Child maltreatment and hypertension in young adulthood. BMC Public Health. 2014 Nov 6;14:1149. doi: 10.1186/1471-2458-14-1149. PMID 25374338
- [Background] Garad Y, Maximova K, MacKinnon N, McGrath JJ, Kozyrskyj AL, Colman I. Sex-Specific Differences in the Association Between Childhood Adversity and Cardiovascular Disease in Adulthood: Evidence From a National Cohort Study. Can J Cardiol. 2017 Aug;33(8):1013-1019. doi: 10.1016/j.cjca.2017.05.008. Epub 2017 May 19. PMID 28754386
- [Background] Murphy MO, Herald JB, Leachman J, Villasante Tezanos A, Cohn DM, Loria AS. A model of neglect during postnatal life heightens obesity-induced hypertension and is linked to a greater metabolic compromise in female mice. Int J Obes (Lond). 2018 Jul;42(7):1354-1365. doi: 10.1038/s41366-018-0035-z. Epub 2018 Feb 23. PMID 29535450
- [Background] Wainstock T, Shoham-Vardi I, Glasser S, Anteby E, Lerner-Geva L. Fetal sex modifies effects of prenatal stress exposure and adverse birth outcomes. Stress. 2015 Jan;18(1):49-56. doi: 10.3109/10253890.2014.974153. Epub 2014 Dec 29. PMID 25319674
- [Background] Barrett ES, Swan SH. Stress and Androgen Activity During Fetal Development. Endocrinology. 2015 Oct;156(10):3435-41. doi: 10.1210/en.2015-1335. Epub 2015 Aug 4. PMID 26241065
- [Background] Shiozaki A, Matsuda Y, Satoh S, Saito S. Impact of fetal sex in pregnancy-induced hypertension and preeclampsia in Japan. J Reprod Immunol. 2011 May;89(2):133-9. doi: 10.1016/j.jri.2010.12.011. Epub 2011 Apr 22. PMID 21514961
- [Background] Taylor BD, Ness RB, Klebanoff MA, Tang G, Roberts JM, Hougaard DM, Skogstrand K, Haggerty CL. The impact of female fetal sex on preeclampsia and the maternal immune milieu. Pregnancy Hypertens. 2018 Apr;12:53-57. doi: 10.1016/j.preghy.2018.02.009. Epub 2018 Feb 24. PMID 29674199
- [Background] Jaskolka D, Retnakaran R, Zinman B, Kramer CK. Fetal sex and maternal risk of pre-eclampsia/eclampsia: a systematic review and meta-analysis. BJOG. 2017 Mar;124(4):553-560. doi: 10.1111/1471-0528.14163. Epub 2016 Jun 17. PMID 27315789
- [Background] Valdiviezo C, Garovic VD, Ouyang P. Preeclampsia and hypertensive disease in pregnancy: their contributions to cardiovascular risk. Clin Cardiol. 2012 Mar;35(3):160-5. doi: 10.1002/clc.21965. PMID 22389120
- [Background] Davis EF, Lazdam M, Lewandowski AJ, Worton SA, Kelly B, Kenworthy Y, Adwani S, Wilkinson AR, McCormick K, Sargent I, Redman C, Leeson P. Cardiovascular risk factors in children and young adults born to preeclamptic pregnancies: a systematic review. Pediatrics. 2012 Jun;129(6):e1552-61. doi: 10.1542/peds.2011-3093. Epub 2012 May 21. PMID 22614768
- [Background] Daniels SR, Pratt CA, Hayman LL. Reduction of risk for cardiovascular disease in children and adolescents. Circulation. 2011 Oct 11;124(15):1673-86. doi: 10.1161/CIRCULATIONAHA.110.016170. No abstract available. PMID 21986774
- [Background] Daniels SR, Pratt CA, Hollister EB, Labarthe D, Cohen DA, Walker JR, Beech BM, Balagopal PB, Beebe DW, Gillman MW, Goodrich JM, Jaquish C, Kit B, Miller AL, Olds D, Oken E, Rajakumar K, Sherwood NE, Spruijt-Metz D, Steinberger J, Suglia SF, Teitelbaum SL, Urbina EM, Van Horn L, Ward D, Young ME. Promoting Cardiovascular Health in Early Childhood and Transitions in Childhood through Adolescence: A Workshop Report. J Pediatr. 2019 Jun;209:240-251.e1. doi: 10.1016/j.jpeds.2019.01.042. Epub 2019 Mar 20. No abstract available. PMID 30904171
- [Background] Van Buren DJ, Tibbs TL. Lifestyle interventions to reduce diabetes and cardiovascular disease risk among children. Curr Diab Rep. 2014 Dec;14(12):557. doi: 10.1007/s11892-014-0557-2. PMID 25344792
- [Background] Sung-Chan P, Sung YW, Zhao X, Brownson RC. Family-based models for childhood-obesity intervention: a systematic review of randomized controlled trials. Obes Rev. 2013 Apr;14(4):265-78. doi: 10.1111/obr.12000. Epub 2012 Nov 9. PMID 23136914
- [Background] Loveman E, Al-Khudairy L, Johnson RE, Robertson W, Colquitt JL, Mead EL, Ells LJ, Metzendorf MI, Rees K. Parent-only interventions for childhood overweight or obesity in children aged 5 to 11 years. Cochrane Database Syst Rev. 2015 Dec 21;2015(12):CD012008. doi: 10.1002/14651858.CD012008. PMID 26690844
- [Background] Campbell F, Conti G, Heckman JJ, Moon SH, Pinto R, Pungello E, Pan Y. Early childhood investments substantially boost adult health. Science. 2014 Mar 28;343(6178):1478-85. doi: 10.1126/science.1248429. PMID 24675955
- [Background] Brody GH, Yu T, Miller GE, Ehrlich KB, Chen E. Preventive parenting intervention during childhood and young black adults' unhealthful behaviors: a randomized controlled trial. J Child Psychol Psychiatry. 2019 Jan;60(1):63-71. doi: 10.1111/jcpp.12968. Epub 2018 Sep 11. PMID 30203840
- [Background] Olds DL. Prenatal and infancy home visiting by nurses: from randomized trials to community replication. Prev Sci. 2002 Sep;3(3):153-72. doi: 10.1023/a:1019990432161. PMID 12387552
- [Background] Olds DL, Henderson CR Jr, Tatelbaum R, Chamberlin R. Improving the delivery of prenatal care and outcomes of pregnancy: a randomized trial of nurse home visitation. Pediatrics. 1986 Jan;77(1):16-28. PMID 3510017
- [Background] Olds DL, Henderson CR Jr, Chamberlin R, Tatelbaum R. Preventing child abuse and neglect: a randomized trial of nurse home visitation. Pediatrics. 1986 Jul;78(1):65-78. PMID 2425334
- [Background] Olds DL, Eckenrode J, Henderson CR Jr, Kitzman H, Powers J, Cole R, Sidora K, Morris P, Pettitt LM, Luckey D. Long-term effects of home visitation on maternal life course and child abuse and neglect. Fifteen-year follow-up of a randomized trial. JAMA. 1997 Aug 27;278(8):637-43. PMID 9272895
- [Background] Olds D, Henderson CR Jr, Cole R, Eckenrode J, Kitzman H, Luckey D, Pettitt L, Sidora K, Morris P, Powers J. Long-term effects of nurse home visitation on children's criminal and antisocial behavior: 15-year follow-up of a randomized controlled trial. JAMA. 1998 Oct 14;280(14):1238-44. doi: 10.1001/jama.280.14.1238. PMID 9786373
- [Background] Eckenrode J, Campa M, Luckey DW, Henderson CR Jr, Cole R, Kitzman H, Anson E, Sidora-Arcoleo K, Powers J, Olds D. Long-term effects of prenatal and infancy nurse home visitation on the life course of youths: 19-year follow-up of a randomized trial. Arch Pediatr Adolesc Med. 2010 Jan;164(1):9-15. doi: 10.1001/archpediatrics.2009.240. PMID 20048236
- [Background] Kitzman H, Olds DL, Henderson CR Jr, Hanks C, Cole R, Tatelbaum R, McConnochie KM, Sidora K, Luckey DW, Shaver D, Engelhardt K, James D, Barnard K. Effect of prenatal and infancy home visitation by nurses on pregnancy outcomes, childhood injuries, and repeated childbearing. A randomized controlled trial. JAMA. 1997 Aug 27;278(8):644-52. PMID 9272896
- [Background] Kitzman H, Olds DL, Sidora K, Henderson CR Jr, Hanks C, Cole R, Luckey DW, Bondy J, Cole K, Glazner J. Enduring effects of nurse home visitation on maternal life course: a 3-year follow-up of a randomized trial. JAMA. 2000 Apr 19;283(15):1983-9. doi: 10.1001/jama.283.15.1983. PMID 10789666
- [Background] Olds DL, Kitzman H, Cole R, Robinson J, Sidora K, Luckey DW, Henderson CR Jr, Hanks C, Bondy J, Holmberg J. Effects of nurse home-visiting on maternal life course and child development: age 6 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1550-9. doi: 10.1542/peds.2004-0962. PMID 15574614
- [Background] Olds DL, Kitzman H, Hanks C, Cole R, Anson E, Sidora-Arcoleo K, Luckey DW, Henderson CR Jr, Holmberg J, Tutt RA, Stevenson AJ, Bondy J. Effects of nurse home visiting on maternal and child functioning: age-9 follow-up of a randomized trial. Pediatrics. 2007 Oct;120(4):e832-45. doi: 10.1542/peds.2006-2111. PMID 17908740
- [Background] Kitzman HJ, Olds DL, Cole RE, Hanks CA, Anson EA, Arcoleo KJ, Luckey DW, Knudtson MD, Henderson CR Jr, Holmberg JR. Enduring effects of prenatal and infancy home visiting by nurses on children: follow-up of a randomized trial among children at age 12 years. Arch Pediatr Adolesc Med. 2010 May;164(5):412-8. doi: 10.1001/archpediatrics.2010.76. PMID 20439791
- [Background] Olds DL, Kitzman HJ, Cole RE, Hanks CA, Arcoleo KJ, Anson EA, Luckey DW, Knudtson MD, Henderson CR Jr, Bondy J, Stevenson AJ. Enduring effects of prenatal and infancy home visiting by nurses on maternal life course and government spending: follow-up of a randomized trial among children at age 12 years. Arch Pediatr Adolesc Med. 2010 May;164(5):419-24. doi: 10.1001/archpediatrics.2010.49. PMID 20439792
- [Background] Olds DL, Kitzman H, Knudtson MD, Anson E, Smith JA, Cole R. Effect of home visiting by nurses on maternal and child mortality: results of a 2-decade follow-up of a randomized clinical trial. JAMA Pediatr. 2014 Sep;168(9):800-6. doi: 10.1001/jamapediatrics.2014.472. PMID 25003802
- [Background] Conti G, Kitzman H, Smith JA, Olds DL. Effects of prenatal/Infancy home visiting on maternal and offspring obesity and blood pressure through age 18. In preparation.
- [Background] Olds DL, Robinson J, O'Brien R, Luckey DW, Pettitt LM, Henderson CR Jr, Ng RK, Sheff KL, Korfmacher J, Hiatt S, Talmi A. Home visiting by paraprofessionals and by nurses: a randomized, controlled trial. Pediatrics. 2002 Sep;110(3):486-96. doi: 10.1542/peds.110.3.486. PMID 12205249
- [Background] Olds DL, Robinson J, Pettitt L, Luckey DW, Holmberg J, Ng RK, Isacks K, Sheff K, Henderson CR Jr. Effects of home visits by paraprofessionals and by nurses: age 4 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1560-8. doi: 10.1542/peds.2004-0961. PMID 15574615
- [Background] Olds DL, Holmberg JR, Donelan-McCall N, Luckey DW, Knudtson MD, Robinson J. Effects of home visits by paraprofessionals and by nurses on children: follow-up of a randomized trial at ages 6 and 9 years. JAMA Pediatr. 2014 Feb;168(2):114-21. doi: 10.1001/jamapediatrics.2013.3817. PMID 24296904
- [Background] Grundy E, Kravdal O. Do short birth intervals have long-term implications for parental health? Results from analyses of complete cohort Norwegian register data. J Epidemiol Community Health. 2014 Oct;68(10):958-64. doi: 10.1136/jech-2014-204191. Epub 2014 Jul 9. PMID 25009153
- [Background] Khatiwada S, Rajendra KC, Gautam S, Lamsal M, Baral N. Thyroid dysfunction and dyslipidemia in chronic kidney disease patients. BMC Endocr Disord. 2015 Oct 29;15:65. doi: 10.1186/s12902-015-0063-9. PMID 26510920
- [Background] Lawlor DA, Davey Smith G, Whincup P, Wannamethee G, Papacosta O, Dhanjil S, Griffin M, Nicolaides AN, Ebrahim S. Association between offspring birth weight and atherosclerosis in middle aged men and women: British Regional Heart Study. J Epidemiol Community Health. 2003 Jun;57(6):462-3. doi: 10.1136/jech.57.6.462. No abstract available. PMID 12775796
- [Background] Lawlor DA, Davey Smith G, Ebrahim S. Birth weight of offspring and insulin resistance in late adulthood: cross sectional survey. BMJ. 2002 Aug 17;325(7360):359. doi: 10.1136/bmj.325.7360.359. PMID 12183306
- [Background] Cronk L. Preferential parental investment in daughters over sons. Hum Nat. 1991 Dec;2(4):387-417. doi: 10.1007/BF02692198. PMID 24222341
- [Background] Cronk, L. Parental Favoritism toward Daughters. Am Sci. 1993;81(3):272-279.
- [Background] Hopcroft, R. Parental status and differential investment in sons and daughters: Trivers-Willard Revisited. Soc Forces. 2005;83(3):1111-1136.
- [Background] Gibson MA. Does Investment in the Sexes Differ When Fathers Are Absent? : Sex-biased Infant Survival and Child Growth in Rural Ethiopia. Hum Nat. 2008 Sep;19(3):263-76. doi: 10.1007/s12110-008-9044-2. PMID 26181617
- [Background] Veloudi P, Sharman JE. Methodological factors affecting quantification of blood pressure variability: a scoping review. J Hypertens. 2018 Apr;36(4):711-719. doi: 10.1097/HJH.0000000000001606. PMID 29176390
- [Background] Lynch BM, Friedenreich CM, Khandwala F, Liu A, Nicholas J, Csizmadi I. Development and testing of a past year measure of sedentary behavior: the SIT-Q. BMC Public Health. 2014 Sep 1;14:899. doi: 10.1186/1471-2458-14-899. PMID 25179551
- [Background] Bull FC, Maslin TS, Armstrong T. Global physical activity questionnaire (GPAQ): nine country reliability and validity study. J Phys Act Health. 2009 Nov;6(6):790-804. doi: 10.1123/jpah.6.6.790. PMID 20101923
- [Background] Subar AF, Thompson FE, Kipnis V, Midthune D, Hurwitz P, McNutt S, McIntosh A, Rosenfeld S. Comparative validation of the Block, Willett, and National Cancer Institute food frequency questionnaires : the Eating at America's Table Study. Am J Epidemiol. 2001 Dec 15;154(12):1089-99. doi: 10.1093/aje/154.12.1089. PMID 11744511
- [Background] Mollayeva T, Thurairajah P, Burton K, Mollayeva S, Shapiro CM, Colantonio A. The Pittsburgh sleep quality index as a screening tool for sleep dysfunction in clinical and non-clinical samples: A systematic review and meta-analysis. Sleep Med Rev. 2016 Feb;25:52-73. doi: 10.1016/j.smrv.2015.01.009. Epub 2015 Feb 17. PMID 26163057
- [Background] Searle SR. Linear models. New York, NY: Wiley;1971.
- [Background] McCullagh P, Nelder JA. Generalized linear models. London, England: Chapman and Hall/CRC;1983
- [Background] Schall R. Estimation in generalized linear models with random effects. Biometrika 1991;78(4):719-27.
- [Background] Russ Wolfinger & Michael O'connell (1993) Generalized linear mixed models a pseudo-likelihood approach, Journal of Statistical Computation and Simulation, 48:3-4, 233-243, DOI: 10.1080/00949659308811554
- [Background] Charles R. Henderson Jr & C.R. Henderson (1979) Analysis of covariance in mixed models with unequal subclass numbers, Communications in Statistics - Theory and Methods, 8:8, 751-787, DOI: 10.1080/03610927908827798
- [Background] Laird NM, Ware JH. Random-effects models for longitudinal data. Biometrics. 1982 Dec;38(4):963-74. PMID 7168798
- [Background] Ruppert D, Wand, MP, Carroll RJ. Semiparametric regression. New York, NY: Cambridge University Press; 2003.
- [Background] Kaplan EL, Meier P. Nonparametric estimation from incomplete observations. J Am Stat Assoc. 1958;53(282):457-481
- [Background] Klein JP. Competing risks. WIREs Comp Stat. 2010;2(3):333-339.
- [Background] Gray RJ. A class of K-sample tests for comparing the cumulative incidence of a competing risk. Ann Stat. 1988;16(3):1141-54.
- [Background] Cox, DR. Regression models and life-tables. J R Stat Soc Series B Stat Methodol. 1972;34(2):187-220.
- [Background] MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychol Methods. 2002 Mar;7(1):83-104. doi: 10.1037/1082-989x.7.1.83. PMID 11928892
- [Background] Bollen KA. Structural equations with latent variables. New York, NY:Wiley;1989.
- [Background] Belloni A, Chernozhukov V, Hansen C. Inference on treatment effects after selection among high-dimensional controls. Rev Econ Stud. 2014;81(2):608-650.
- [Background] Bradley Efron. Trevor Hastie. Iain Johnstone. Robert Tibshirani.
- [Background] MR Osborne, B Presnell, BA Turlach, A new approach to variable selection in least squares problems, IMA Journal of Numerical Analysis, Volume 20, Issue 3, July 2000, Pages 389-403, https://doi.org/10.1093/imanum/20.3.389
- [Background] Little RJA, Rubin DB. Statistical analysis with missing data, 2nd ed. New York, NY:John Wiley and Sons;2002.
- [Background] Olds DL, Kitzman H, Anson E, Smith JA, Knudtson MD, Miller T, Cole R, Hopfer C, Conti G. Prenatal and Infancy Nurse Home Visiting Effects on Mothers: 18-Year Follow-up of a Randomized Trial. Pediatrics. 2019 Dec;144(6):e20183889. doi: 10.1542/peds.2018-3889. Epub 2019 Nov 20. PMID 31748253
- [Background] Cheng, S. The accumulation of (dis)advantage: The intersection of gender and race in the long-term wage effect of marriage. Am Sociol Rev. 2016;81(1):29-56.
- [Background] Waite LJ. Does marriage matter? Demography. 1995 Nov;32(4):483-507. No abstract available. PMID 8925942
- [Background] .Ludwig, V., Brüderl, J. Is there a male marital wage premium? New evidence from the United States. Am Sociol Rev. 2018;83(4):744-770.
- [Background] Barr AB, Culatta E, Simons RL. Romantic relationships and health among African American young adults: linking patterns of relationship quality over time to changes in physical and mental health. J Health Soc Behav. 2013;54(3):369-85. doi: 10.1177/0022146513486652. Epub 2013 May 8. PMID 23657713

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT06160037/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT06160037/ICF_001.pdf